CLINICAL TRIAL: NCT03248024
Title: Etude Des Facteurs Explicatifs Des Coûts de la Prise En Charge Des Patients Adultes Atteints d'Une MICI Suivis au CHRU de Nancy et traités Par biothérapie
Brief Title: An Explanatory Factors Analysis of Inflammatory Bowel Diseases(IBD's) Management Costs for Adults Patients Treated by Biotherapy and Followed at Nancy University Hospital
Acronym: FECPEC MICI
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: HEVA - Lyon (Unknown)
Responsible Party: Sponsor
Other Study IDs: FECPEC MICI
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Chronic Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Chronic Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to analyze the factors influencing the medical and non-medical direct costs of patients treated with biotherapy during the last twelve months (infliximab or adalimumab), including biosimilars (infliximab biosimilars: Inflectra ™ and Remsima ™) for treating Crohn's desease or ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

1. Patients consulted at the Gastroenterology services of Nancy University Hospital during the period of inclusion
2. Patients over 18 of age the day of consultation
3. Patients treated at least one time by biotherapy during the last 12 months preceeding inclusion
4. Patients with crohn's disease or ulcerative colitis.
5. Patients accepting to respond to the questionnary

Exclusion Criteria:

* Age under 18 years , the day of consultation
* Patient that not accept or unable to complete the retrospective questionnary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received biotherapy during the last 12 months preceeding consultation for treatment of crohn's disease or ulcerative colitis.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Retrospective health care consumption | one year
  Desease treatment cost individual level data